CLINICAL TRIAL: NCT06617039
Title: The Impact of Low-Dose Esketamine Combined With Ciprofol on the Quality of Early Postoperative Recovery Among Elderly Patients Undergoing Painless Gastroscopy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Jiangsu People's Hospital (Other)
Responsible Party: Principal Investigator, Ju Gao, Study Director, Northern Jiangsu People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024ky251
Record Dates: First submitted 2024-09-20; First posted 2024-09-27 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Quality of Postoperative Recovery
MeSH Terms: interventions — Remifentanil; (2-(1R)-1-cyclopropyl)ethyl-6-isopropyl-phenol; Esketamine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Ciprofol group (C group) (Active Comparator): Ciprofol group will be started with ciprofol 0.2-0.4 mg/kg.
  Interventions: Drug: Ciprofol
- The group of remifentanil 0.5ug/kg combined with ciprofol(R group) (Experimental): R group will be started with remifentanil 0.5ug/kg and ciprofol 0.2-0.4 mg/kg.
  Interventions: Drug: Remifentanil and ciprofol
- The group of esketamine 0.3mg/kg combined with ciprofol(E1 group) (Experimental): E1 group will be started with esketamine 0.3mg/kg and ciprofol 0.2-0.4 mg/kg.
  Interventions: Drug: esketamine 0.3mg/kg and ciprofol
- The group of esketamine 0.5mg/kg combined with ciprofol(E2 group) (Experimental): E2 group will be started with esketamine 0.5mg/kg and ciprofol 0.2-0.4 mg/kg.
  Interventions: Drug: esketamine 0.5mg/kg and ciprofol

INTERVENTIONS:
Drug: Remifentanil and ciprofol — R group will be started with remifentanil 0.5ug/kg and ciprofol 0.4 mg/kg.
  Arms: The group of remifentanil 0.5ug/kg combined with ciprofol(R group)
Drug: esketamine 0.3mg/kg and ciprofol — Anesthesia induction was initiated by esketamine 0.3mg/kg, followed by ciprofol 0.2-0.4mg/kg.
  Arms: The group of esketamine 0.3mg/kg combined with ciprofol(E1 group)
Drug: esketamine 0.5mg/kg and ciprofol — Anesthesia induction was initiated by esketamine 0.5mg/kg, followed by ciprofol 0.2-0.4mg/kg.
  Arms: The group of esketamine 0.5mg/kg combined with ciprofol(E2 group)
Drug: Ciprofol — Ciprofol group will be started with ciprofol 0.2-0.4 mg/kg.
  Arms: Ciprofol group (C group)

SUMMARY:
To explore the impact of esketamine combined with ciprofol on the quality of early postoperative recovery in elderly patients undergoing painless gastroscopy, as well as the effectiveness and safety of this regimen.

ELIGIBILITY:
Inclusion Criteria:

* 1. Scheduled painless gastroscopy examination and treatment

  2. Age 60-75 years old

  3. ASA grade Ⅰ-Ⅱ

  4. The respiratory tract is unobstructed and there is no difficult airway

  5. No history of allergy to etomidate and cyclopropofol

  6. Participants with normal heart, liver, lung, and kidney functions

  7. Able to complete the QoR-15, MMSE, and HADS scale assessments

  8. lnformed consent, voluntary participation in the trial, and signed by the patient informed consent

Exclusion Criteria:

* 1. Participants with concurrent dysfunction of major organs.

  2. Participants with a history of mental illness and abuse of sedative drugs

  3. Participants with allergies or contraindications to the study drugs

  4. Participants with severe visual, auditory, or speech communication impairments

  5. Participants with acute gastrointestinal inflammation or obstruction

  6. History of uncontrolled diabetes, hypertension, and hypotension

  7. Participants with malignant tumors, severe hyperkalemia, bronchial asthma, or excessive obesity (BMI > 30kg/m2)

  8. Participants with aneurysmal vascular diseases of the thoracic and abdominal aorta, intracranial and peripheral arterial vessels.

  9. Unable to cooperate with the QoR-15, MMSE, and HADS scale assessments

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 376 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
postoperative day 1(POD1) Quality of Recovery(QoR)-15 questionnaire score | Baseline (30 min before surgery), postoperative day 1
  Quality of life will be evaluated using Quality of Recovery(QoR)-15 questionnaire score at postoperative day 1(minimum value : 0, maximum value : 150, the higher the score, the better the result)

SECONDARY OUTCOMES:
postoperative day 3(POD3) Quality of Recovery(QoR)-15 questionnaire score | Postoperative day 3 and 7
  Quality of life will be evaluated using Quality of Recovery(QoR)-15 questionnaire score at postoperative day 3(minimum value : 0, maximum value : 150, the higher the score, the better the result)
Cognitive function assessment | Baseline (30 min before surgery), postoperative day 1,3 and 7
  A Mini-Mental State Examination (MMSE) is a set of 11 questions that doctors and other healthcare professionals commonly use to check for cognitive impairment (problems with thinking, communication, understanding and memory). MMSE has a maximum total score of 30, with higher scores manifesting a better cognitive performance.
Hospital anxiety and depression scale ( HADS ) score. | Baseline (30 min before surgery), postoperative day 1,3 and 7
  Postoperative anxiety and depression scores will be measured by the Hospital Anxiety and Depression Scale, on the morning(8-10 am) of postoperative days (PODs) 1,3 and 7 , a score of 8 points or higher will be diagnosed as depression or anxiety.
Dosage of ciprofol | During endoscopic examination
  Consumption of ciprofol during endoscopic examination
Heart rate (HR) | Baseline，during surgery and arrived at PACU (up to 30 minutes after surgery)
  Throughout the procedure, the heart rate (HR) was continuously monitored.
Pulse oxygen saturation (SpO2) | Baseline, during surgery and arrived at PACU (up to 30 minutes after surgery)
  Throughout the procedure, the pulse oxygen saturation (SpO2) were continuously monitored.
Mean blood pressure (MBP) | Baseline, during surgery and arrived at PACU (up to 30 minutes after surgery)
  Throughout the procedure, the mean blood pressure (MBP) was measured at 1-minute intervals.
Patient satisfaction levels | 30 minutes at recovery room.
  The patients express their satisfaction with procedures on a visual analogue score, ranging from 0 to 10, where 0 is the minimum and 10 is the maximum satisfaction level.

OTHER OUTCOMES:
The incidence of all drug-related adverse events | Within 72hours after surgery
  All drug-related adverse events including bradycardia, hypotension, tachycardia, hypertension, arrhythmia, nystagmus, hypersalivation, euphoria, emergence agitation, hallucinations, dreaminess and nightmares during surgery or before discharge.etc.Patients will be followed up for 3 days consecutively(at 8-10am).

CONTACTS AND LOCATIONS:
Locations (1):
- Subei People's Hospital of Jiangsu Province, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No